CLINICAL TRIAL: NCT00143533
Title: Phase I Study of Intravenous Irinotecan Using Selective Gastrointestinal Decontamination for Prevention of Diarrhea in Relapsed or Refractory Pediatric Solid Tumors
Brief Title: Prevention of Diarrhea in Patients Taking IV Irinotecan for Relapsed or Difficult to Treat Pediatric Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPTCEF
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2011-09

CONDITIONS: Neoplasm; Diarrhea
Keywords: Solid Tumors
MeSH Terms: conditions — Neoplasms; Diarrhea | interventions — Irinotecan; Cefpodoxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Irinotecan, Cefpodoxime

INTERVENTIONS:
Drug: Irinotecan, Cefpodoxime — See Detailed description section for treatment details.

SUMMARY:
The primary purpose of this study is to estimate the maximum tolerated dose of irinotecan with the use of cefpodoxime for pediatric solid tumor patients.

DETAILED DESCRIPTION:
This is a phase I study with the exploratory investigation of at least four dosage levels (20, 30, 45, 60) to define the tolerable dose for phase II studies. Primary consideration will be given to determinations of the qualitative and quantitative toxicity of the administration of irinotecan with cefpodoxime, and pharmacokinetics of irinotecan when given with cefpodoxime.

Standard phase I escalation study in cohorts of 3-6 patients. Starting level is 20 mg/m2/d, and subsequent levels will be 30 mg/m2/d, 45 mg/m2/d and 60 mg/m2/d. An amendment to the study has included an intermediate level at 40 mg/m2/d.

Irinotecan will be administered as a 60-minute intravenous infusion daily for 5 consecutive days, followed by a 2 day rest, and followed by an additional 5 consecutive days course [(qd x 5) x 2]. Twenty-one days from the first dose will be considered one cycle of therapy. Cefpodoxime will be given orally at 10 mg/kg/day divided BID, starting 2 days prior to the beginning of the first course of irinotecan, and will be continued for the duration of study participation.

Additional objectives include:

* To describe the pharmacokinetics of intravenous irinotecan when given with oral cefpodoxime.
* To describe the dose-limiting toxicity/ies of irinotecan given on the [(qd x 5) x 2] with oral cefpodoxime.
* To evaluate the effect of the administration of oral cefpodoxime on the amount of intestinal beta-glucuronidase.
* To correlate the incidence and severity of diarrhea with the amount of intestinal beta-glucuronidase.
* To describe the toxicities of irinotecan given at doses above 20 mg/m2/d
* To note tumor responses within the confines of a phase I trial

ELIGIBILITY:
Inclusion Criteria:

* Subjects under 21 years of age at the time of initial diagnosis
* Recurrent solid tumors that have shown to be unresponsive to conventional treatment for their disease, or subjects with newly diagnosed tumors for whom no conventional treatment is available
* Histologic verification of solid tumor malignancy at original diagnosis
* Adequate performance status
* Neurologic deficits in subjects with central nervous system (CNS) tumors must have been relatively stable for a minimum of 2 weeks prior to study entry
* Subjects must have recovered from the toxic effects of all prior chemotherapy before entering the study
* Adequate bone marrow, renal and hepatic function

Exclusion Criteria:

* No active infection at time of protocol entry, and should not be receiving antibiotics other than P. carinii pneumonia prophylaxis.
* Patients must not be pregnant or lactating.
* Patients must not be taking an enzyme-inducing anticonvulsant (e.g., phenobarbital, phenytoin, or carbamazepine), rifampin, or St. John's Wort. Dexamethasone is not to be used as an antiemetic.
* Patients must not have had any previous allergic reactions to penicillin or cephalosporins.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2003-09; Primary Completion 2010-09 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities | September 2010

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Rodriguez-Galindo, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org